CLINICAL TRIAL: NCT03301259
Title: Evaluation of the Post Treatment Pain After Instrumentation of Root Canals With a Single File Reciprocating (Wave-One Ni Ti File, DENTSPLY Maillefer) or Rotary(One Shape, Micro Mega, France) File System in Patient With Asymptomatic Necrotic Molars
Brief Title: Postoperative Pain Following Treatment of Asymptomatic Necrotic Mandibular Molars in Single Visit Using Wave-one Reciprocating Instruments Versus One-Shape Rotary Instruments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ragab Mohamed, master candidate at endodontic department faculty of oral and dental medicine CU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-06-17
Record Dates: First submitted 2017-09-24; First posted 2017-10-04 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Necrotic Pulp
Keywords: Necrotic pulp; wave-one; one-shape; periapical lesion
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wave -one reciprocating system (Experimental): The reciprocating single file systems WaveOne (Maillefer, Ballaigues, Switzerland) provide more flexibility of the M-wire Ni-Ti alloy, greater resistance to cyclic fatigue and better handling of narrow and curved canals than the traditional Ni-Ti instruments Root canal preparation will be done with theWaveOne System with strict adherence to the manufacturer's instructions. After coronal preflaring with File ISO 21 taper 8% instrument with 2.5% sodium hypochlorite as the irrigant, working length was determined and a glide path will created.
  The Red file R 25 taper 8% will be used for preparing the mesial canal; and the Black ISO 40 taper 8% file will be used for preparing the distal canals where there is only a single canal.
  Interventions: Other: One-shape rotationary system
- OneShape (Experimental): OneShape (MICRO-MEGA) rotary nickel-titanium use roation movement and available in two sizes N°30 - .06 rotary files. , N°25 - .06
  Interventions: Other: One-shape rotationary system

INTERVENTIONS:
Other: One-shape rotationary system — OneShape (MICRO-MEGA) rotary nickel-titanium use roation movement and available in two sizes N°30 - .06 rotary files. , N°25 - .06

SUMMARY:
The aim of this study is to evaluate the post treatment pain after instrumentation of root canals with a single file reciprocating (Wave-One Ni Ti file, DENTSPLY Maillefer) or rotary(One Shape, Micro Mega, France) file system in patient with asymptomatic necrotic molars This trial will help to clinically evaluate the use of reciprocating motion in endodontic treatment in necrotic teeth without periapical lesion therefore reduce the post-obtuation pain

DETAILED DESCRIPTION:
The aim of this study is to evaluate the post treatment pain after instrumentation of root canals with a single file reciprocating (Wave-One Ni Ti file, DENTSPLY Maillefer) or rotary(One Shape, Micro Mega, France) file system in patient with asymptomatic necrotic molars This trial will help to clinically evaluate the use of reciprocating motion in endodontic treatment in necrotic teeth without periapical lesion therefore reduce the post-obtuation pain

Sample

if the success rate (no pain) for wave one subjects is 0.3, we will need to study 17 patients in each group to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.8. the type 1 error probability associated with this test of this null hypothesis. This no is to be increased to total no 42 to compensate for losses during follow up , the sample size was calcukated by the PS program

Patients are recruited for the clinical trial from the clinic of endodontics at the Faculty of Oral and Dental Medicine, Cairo University to meet the target sample size.

A random sequence will be generated by computer software, (http://www.random.org/) in the Center of Evidence Based Dentistry, Cairo University. This table will be kept with a co-investigator

The operator finds an eligible participant, then to assign the Participant to either group according to the generated random sequence.

The operator finds an eligible participant, then to assign the Participant to either group according to the generated random sequence.

We will generate the random sequence, assign the participants to the intervention or control groups.

The operators will enroll the participants after they find the eligible ones.

Outpatients of the clinic of endodontics at the Faculty of Oral and Dental Medicine, Cairo University, Egypt.

* The dental Unit is Adec 200 U.S.A.
* The x-ray Machine is ViVi, S.r.I, Italy
* The x-ray films are Kodac, speed D, size 2 or Digital (RVG)
* The operator is a master degree student in the department of Endodontics

Radiographic examination using periapical radiographic film which shows normal periapical tissues with normal lamina dura and width of the periodontal membrane space and absence of periapical lesion

Assessment of pre-operative pain:

The patients will be asked to record the level of pain on a VAS. The patient will be trained that 0 is no pain, 10 is the worst pain, and he will be asked to estimate the pain from 0 to 10 which then will be scored as follows:

0 No pain. From 1-3 mild pain. From 4-5 moderate pain. From 7-10 severe pain

The standard procedure for both groups in single visit

Standard access cavity will be prepared. Isolation will be performed using rubber dam.

K file 10 or 15 will be used to check the patency of the canal. ENDOFLARE will be used for enlarging the coronal third of the canal in cases which will be treated with One Shape Lubricant gel will be used as a lubricant and 2.5% NaOCl as irrigant. Determination of the working length of canal will be done by electronic apex locator and confirmed by periapical radiograph.

Intervention group Root canal preparation will be done with theWaveOne System with strict adherence to the manufacturer's instructions. After coronal preflaring with File ISO 21 taper 8% instrument with 2.5% sodium hypochlorite as the irrigant, working length was determined and a glide path will created.

The Red file R 25 taper 8% will be used for preparing the mesial canal; and the Black ISO 40 taper 8% file will be used for preparing the distal canals where there is only a single canal.

Control Group: canals will be prepared by OneShape (MICRO-MEGA) rotary nickel-titanium file at 400 rpm. The preparation will be stopped by One Shape N°25 - .06 in mesial canals and distal roots with 2 canals; while in case of a single distal canal, the preparation will be stopped by One Shape apical N°30 - .06 rotary files.

Obturation:

After instrumentation and final irrigation, canals will be dried with paper points.

Teeth will be obturated during the initial appointment using epoxy resin sealer.

All the patients will be asked to take a placebo if they experience pain after the procedures. If the patient experience moderate pain he is allowed to take 50mg diclofenac potassium (cataflam 50mg). Any of the patients with intolerable pain will be requested to visit the clinician for emergency treatment. The patients will be asked to record the no. of pills taken and the time at which it was taken.

Assessment of post-operative pain:

Post-operative pain is defined as any degree of pain that occurs after initiation of root canal treatment, while flare up is defined as the development or continuation of pain and/or swelling after endodontic treatment.

The will be asked to record the level of pain at 6 hours, 24 hours, 48 hours and 7days after obturation.

The patient will be trained that 0 is no pain, 10 is the worst pain that interfere with his daily routine, and he will be asked to estimate the pain as follows:

0 No pain. From 1-3 mild pain. From 4-5 moderate pain. From 7-10 severe pain

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients
2. Patient's age between 25-50 years.
3. Mandibular molars diagnosed clinically as necrotic with normal apical tissues.
4. Positive patient's acceptance for participation in the study.
5. Both genders are included.
6. Patients able to sign informed consent.
7. Normal periodontal tissues.
8. Normal periapical tissues on the radiograph

Exclusion Criteria:

1. Patients with complicating systemic disease.
2. Having severe pain and/or acute apical abscesses.
3. Under the age of 25 years.
4. Patients using antibiotics or analgesic 12 hours before the procedures.
5. Having multiple teeth that required treatment.
6. With non-restorable and/or periodontally compromised teeth.
7. Retreatment cases
8. Presence of sinus tract
9. Pregnancy

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | changes after 6 hours , 24 hours , 48 hours , 7 days The patient will be trained that 0 is no pain, 10 is the worst pain that interfere with his daily routine, and he will be asked to estimate the pain from 0 to 10
  Post operative pain after mechanical preparation with wave one and one shape using VAS scale from 0 to 10
  Post-operative pain is defined as any degree of pain that occurs after initiation of root canal treatment, while flare up is defined as the development or continuation of pain and/or swelling after endodontic treatment.
  The will be asked to record the level of pain at 6 hours, 24 hours, 48 hours and 7days after obturation.
  The patient will be trained that 0 is no pain, 10 is the worst pain that interfere with his daily routine, and he will be asked to estimate the pain as follows:
  0 No pain. From 1-3 mild pain. From 4-5 moderate pain. From 7-10 severe pain

IPD SHARING:
Plan to Share IPD: Undecided